CLINICAL TRIAL: NCT02227459
Title: A Phase 1b/2, Open Label, Randomized, Repeat Dose, Dose Escalation Study to Evaluate the Safety, Tolerability, Biological Activity, and Pharmacokinetics of ND-L02-s0201 Injection, A Vitamin A-coupled Lipid Nanoparticle Containing siRNA Against HSP47, in Subjects With Moderate to Extensive Hepatic Fibrosis (METAVIR F3-4)
Brief Title: Phase 1b/2, Open Label, Repeat Dose, Dose Escalation Study of ND-L02-s0201 Injection in Subjects With Moderate to Extensive Fibrosis (METAVIR F3-4)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Nitto Denko Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ND-L02-s0201-002
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Moderate to Extensive Hepatic Fibrosis (METAVIR F3-4)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: Arm A (Experimental): Once a week dosing
  Interventions: Drug: ND-L02-s0201 Injection
- Experimental: Arm B (Experimental): Twice a week dosing
  Interventions: Drug: ND-L02-s0201 Injection

INTERVENTIONS:
Drug: ND-L02-s0201 Injection
  Other Names: BMS-986263

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of multiple doses of ND-L02-s0201 in subjects with moderate to extensive hepatic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 75 years
2. Diagnosis of METAVIR F3-4 hepatic fibrosis determined by liver biopsy done within 12 months before screening (Cohort 1) or at the pre-dose biopsy within 6 weeks before treatment (Cohorts 2 and 3)
3. Adequate and stable synthetic hepatic function (albumin ≥ 3 g/dL, international normalized ratio [INR] ≤ 1.4 x upper limit of normal [ULN] and stable by prior medical history).
4. Adequate and stable hepatic function as measured by alkaline phosphatase (ALP), alanine transaminase (ALT), aspartate transaminase (AST), gamma glutamate transferase (GGTP), and total bilirubin (ALT/AST ≤ 5 x ULN, ALP ≤ 4 x ULN, GGTP ≤ 4 x ULN, bilirubin ≤ 2x ULN and stable by prior medical history).
5. Platelet count ≥ 75,000/mm3, hemoglobin ≥ 10 g/dL, and white blood cell count (WBC) > 3000/µL.
6. No signs of decompensated liver disease (ascites, hepatic encephalopathy, or variceal bleeding).
7. No clinically significant abnormalities on 12-lead electrocardiogram (ECG).
8. No other intercurrent medical conditions or infections considered clinically significant by the Investigator.
9. Clinical laboratory assessments are within the laboratory limits of normal values or not considered clinically significant by the Investigator.
10. Vitamin A levels at screening must be less than or equal to the upper limit of normal (ULN 95 µg/dL or 3.32 µmol/L).
11. Any male subject, if sexually active, agrees to use barrier contraceptive techniques as defined in the protocol. If female, the subject must be of non-childbearing potential as defined in the protocol.
12. Subjects who are active substances abusers may be enrolled at the discretion of the Principal Investigator.
13. Willing and able to provide written informed consent and comply with the study procedures and visit schedule, including follow up visits.

Exclusion Criteria:

1. Any disease or condition which, in the opinion of the Investigator, might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, skeletal, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism, or excretion of ND L02 s0201, or would place the subject at increased risk.
2. On ongoing therapy for HCV/HBV, or received therapy for HCV/HBV within 12 weeks prior to administration of study drug.
3. On interferon therapy for any disease or received interferon therapy for any disease within 12 weeks prior to administration of study drug.
4. History of bone disease, including osteoporosis and osteomalacia, Paget's disease of bone, or a history of unexplained fractures or fractures after minimal trauma.
5. Alpha-fetoprotein (AFP) ≥ 50 ng/mL or signs of abnormality or hepatocellular carcinoma on ultrasound survey of the liver.
6. Carcinoembryonic antigen (CEA) levels above the ULN.
7. Laboratory test results include abnormal values considered to be clinically significant by the Investigator.
8. Participated in a concurrent interventional study with the last intervention occurring within 12 weeks prior to administration of study drug.
9. Taken vitamin A or vitamin D supplements or multi-vitamins that contain vitamin A or vitamin D between the screening visit and administration of study drug.
10. History, within the last 2 years, of alcohol abuse, significant mental illness, or physical dependence on any opioid.
11. Veins unsuitable for repeated venipuncture or IV infusion (eg, veins that are difficult to locate, access or puncture; veins with a tendency to rupture during or after puncture).
12. Received recent treatment with alternative therapies, which, in the opinion of the Investigator, could potentially confound clinical or laboratory assessments.
13. Lost more than 500 mL of blood within 56 days prior to administration of study drug.
14. Body mass index (BMI) > 38 kg/m2.
15. History of human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome-related illness (AIDS).
16. History of malignancy within the last 5 years with the exception of basal cell carcinoma.
17. Woman of childbearing potential.
18. History of hypersensitivity to H2-receptor antagonists.
19. Any other reason that, in the opinion of the Investigator or the Sponsor's Medical Monitor, makes the subject unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with serious and non-serious adverse events | After treatment for 5 consecutive weeks and follow-up through week 24

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lawitz, MD, Principal Investigator — Texas Liver Institute; Rozalina Balabanska, MD, Principal Investigator — Tokuda Hospital
Locations (2):
- Texas Liver Institute, Austin, Texas, United States
- Tokuda Hospital, Sofia, Bulgaria